CLINICAL TRIAL: NCT03532256
Title: Using Text-messaging to Engage Patients and Crowdsource Data: an Opioid Pilot Study
Brief Title: Post-op Crowd Sourcing Health Data Via Text-messaging
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: 827461; HHSF223201810209C (Other: FDA)
Record Dates: First submitted 2018-04-16; First posted 2018-05-22 (Actual); Results first posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: Orthopedic Surgery; Opioid Use; Acute Injuries Knee; Neurosurgery; Surgery
Keywords: Quality Improvement; Prescription Use; Patient Experience; SMS Messaging; Crowd Sourcing
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Treated Patients: This prospective, observational study includes adult patients (age ≥18) undergoing elective surgical procedures within the departments of orthopedics, sports medicine, and neurosurgery, as well as patients treated for an acute injury and prescribed an opioid from the ED who own a mobile phone and can receive SMS text messaging at the University of Pennsylvania or Penn Presbyterian Medical Center.
  Interventions: Behavioral: Observation
- Treated patients randomized to receive survey: A subset of patients (described above) will receive an automated SMS text message with a link to an online survey. This survey contains the script questions about pain management and opioid use.
  Interventions: Behavioral: Observation; Behavioral: Text to online survey
- Treated patients randomized to receive text script: A subset of patients (described above) will receive an automated questionnaire conducted via text message. Questions will be about pain management and opioid use.
  Interventions: Behavioral: Observation; Behavioral: Bi-directional text script

INTERVENTIONS:
Behavioral: Observation — Patients will be contacted postoperatively via an automated text-message to assess pain, functional status, and opioid consumption.
Behavioral: Text to online survey — Subset of surgical patients will receive an automated text message with a link to a secure online survey with questions that assess pain, functional status, and opioid consumption.
  Groups: Treated patients randomized to receive survey
Behavioral: Bi-directional text script — Subset of surgical patients will receive an automated bi-directional text message script with questions that assess pain, functional status, and opioid consumption.
  Groups: Treated patients randomized to receive text script

SUMMARY:
The Center for Disease Control has labeled the opioid prescription drug crisis an "epidemic" in the United States and recently this epidemic has been named a public health emergency. Various medical and surgical societies have begun to release general opioid prescribing guidelines for providers addressing acute pain, but these do not highlight the patient perspective or experience. Identifying an acceptable opioid dose and duration has remained a challenge and is a nuanced process. Though policy and provider driven changes may begin to augment practice, these avenues may miss a crucial perspective; the patient's.

DETAILED DESCRIPTION:
This is a quality improvement project aimed at building upon prior telephone-based patient follow-up. The research team will be launching a text messaging interface to collect and describe patient pain, functional status, and opioid usage with patients undergoing elective surgical procedures within the departments of orthopaedics and sports medicine, as well as patients treated in neurosurgery, general surgery, and the ED who own a mobile phone and can receive SMS text messaging (as measured by pain scale, patient reported functional status, and proportion of opioids used). Additionally, this project aims to evaluate the current standard of care of prescribing opioids to patients among orthopedic surgeons and emergency medicine providers for acute pain.

BACKGROUND

The study team has shown the ability of gathering patient level data from telephone follow up to guide physician behavior. In recent work, providing orthopaedic surgeons with data on patients' unused prescribed opioids has changed practice - patients now reporting a change from twenty unused pills down to seven unused pills.

Though effective, telephone follow up is laborious and time consuming. The researchers seek to test an alternative approach for a rapid, scalable means of engaging patients and gathering patient level data to help inform provider practice.

Text messaging offers a unique opportunity to quickly capture, analyze, and understand the patient experience. The research team has demonstrated the successes of communicating with patients via text-messaging by guiding patients through pre- and postoperative recovery via the program "Engaged Recovery at Penn" (ERAP). This program has enrolled over 900 patients across surgical specialties with automated text-based reminders. The researchers will investigate the intersection of digital patient centered communication, acute pain, and consumption of prescribed opioids to ultimately help inform providers and health systems.

METHODS

The study team will contact adult patients (age ≥18) undergoing elective surgical procedures within the departments of orthopaedics, sports medicine, and neurosurgery, as well as patients undergoing procedures in general surgery and the ED who own a mobile phone and can receive SMS text messaging at the University of Pennsylvania or Penn Presbyterian Medical Center. The researchers will build upon previous work by Dr. Delgado in which patients were approached for follow up data collection via telephone communication and translate the telephone script into a functional and approachable text messaging script. The researchers will work to build an automated bi-directional text script hosted on a secure web portal. The research team will test the ability to engage patients in these departments, gather data, and measure satisfaction with the automated text-messaging system.

Data collected through the online texting portal will be used to demonstrate the ability of bi-directional texting to enhance data collection and then the researchers will utilize this data to develop, implement, and evaluate the use of EMR defaults for opioid prescribing for specific surgical procedures or acute painful conditions.

In addition, the study team will build and deploy an online survey containing the script questions in order to test an alternative to capturing patient data. Using block randomization, a subset of patients will receive either 1) a link to the online survey or 2) the bidirectional text messing script. Patient questions will not change but the method of data collection will test which approach yields a higher response rate. The study team will collect both response and completion rates and evaluate which data collection method is more effective for gathering data using an automated system. Insights gained from this comparison will be used to develop the automated text system and methodology.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 or older
* Undergoing elective surgical procedures within the departments of orthopedics, sports medicine, and neurosurgery, as well as patients undergoing procedures in general surgery and the ED at University of Pennsylvania Hospital or Penn Presbyterian Medical Center
* Own a mobile phone and can receive SMS text messaging

Exclusion Criteria

* Under 18
* Does not own mobile phone
* Owns mobile phone but cannot reliably receive SMS text messages

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (age ≥18) undergoing elective surgical procedures within the departments of orthopedics, sports medicine, and neurosurgery, as well as patients undergoing procedures in general surgery and the ED who own a mobile phone and can receive SMS text messaging at the University of Pennsylvania or Penn Presbyterian Medical Center.
Sampling Method: Non-Probability Sample
Enrollment: 127 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2019-09-16 (Actual); Study Completion 2019-09-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: M. Kit Delgado, MD, MS, Principal Investigator — University of Pennsylvania; Zarina Ali, MD, Principal Investigator — University of Pennsylvania; Anish Agarwal, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared.

REFERENCES:
- [Background] Understanding the Epidemic | Drug Overdose | CDC Injury Center [Internet]. 2017 [cited 2017 Nov 2];Available from: https://www.cdc.gov/drugoverdose/epidemic/index.html
- [Background] Rudd RA, Seth P, David F, Scholl L. Increases in Drug and Opioid-Involved Overdose Deaths - United States, 2010-2015. MMWR Morb Mortal Wkly Rep. 2016 Dec 30;65(50-51):1445-1452. doi: 10.15585/mmwr.mm655051e1. PMID 28033313
- [Background] Compressed Mortality, 1999-2015 Request Form [Internet]. [cited 2017 Nov 2];Available from: https://wonder.cdc.gov/controller/datarequest/D132
- [Background] Pletcher MJ, Kertesz SG, Kohn MA, Gonzales R. Trends in opioid prescribing by race/ethnicity for patients seeking care in US emergency departments. JAMA. 2008 Jan 2;299(1):70-8. doi: 10.1001/jama.2007.64. PMID 18167408
- [Background] Levy B, Paulozzi L, Mack KA, Jones CM. Trends in Opioid Analgesic-Prescribing Rates by Specialty, U.S., 2007-2012. Am J Prev Med. 2015 Sep;49(3):409-13. doi: 10.1016/j.amepre.2015.02.020. Epub 2015 Apr 18. PMID 25896191
- [Background] Manchikanti L, Abdi S, Atluri S, Balog CC, Benyamin RM, Boswell MV, Brown KR, Bruel BM, Bryce DA, Burks PA, Burton AW, Calodney AK, Caraway DL, Cash KA, Christo PJ, Damron KS, Datta S, Deer TR, Diwan S, Eriator I, Falco FJ, Fellows B, Geffert S, Gharibo CG, Glaser SE, Grider JS, Hameed H, Hameed M, Hansen H, Harned ME, Hayek SM, Helm S 2nd, Hirsch JA, Janata JW, Kaye AD, Kaye AM, Kloth DS, Koyyalagunta D, Lee M, Malla Y, Manchikanti KN, McManus CD, Pampati V, Parr AT, Pasupuleti R, Patel VB, Sehgal N, Silverman SM, Singh V, Smith HS, Snook LT, Solanki DR, Tracy DH, Vallejo R, Wargo BW; American Society of Interventional Pain Physicians. American Society of Interventional Pain Physicians (ASIPP) guidelines for responsible opioid prescribing in chronic non-cancer pain: Part 2--guidance. Pain Physician. 2012 Jul;15(3 Suppl):S67-116. PMID 22786449
- [Background] Nicholson B. Responsible prescribing of opioids for the management of chronic pain. Drugs. 2003;63(1):17-32. doi: 10.2165/00003495-200363010-00002. PMID 12487620
- [Background] Gordon AL, Connolly SL. Treating Pain in an Established Patient: Sifting Through the Guidelines. R I Med J (2013). 2017 Oct 2;100(10):41-44. PMID 28968622
- [Background] Dowell D, Haegerich TM, Chou R. CDC Guideline for Prescribing Opioids for Chronic Pain - United States, 2016. MMWR Recomm Rep. 2016 Mar 18;65(1):1-49. doi: 10.15585/mmwr.rr6501e1. PMID 26987082
- [Background] American Academy of Pain Medicine - State Legislative Updates [Internet]. [cited 2017 Nov 2];Available from: http://www.painmed.org/advocacy/state-updates/
- [Background] Preventing Opioid Misuse: Legislative Trends and Predictions > National Conference of State Legislatures [Internet]. [cited 2017 Nov 2];Available from: http://www.ncsl.org/blog/2017/01/31/preventing-opioid-misuse-legislative-trends-and-predictions.aspx
- [Derived] Agarwal AK, Ali ZS, Shofer F, Xiong R, Hemmons J, Spencer E, Abdel-Rahman D, Sennett B, Delgado MK. Testing Digital Methods of Patient-Reported Outcomes Data Collection: Prospective Cluster Randomized Trial to Test SMS Text Messaging and Mobile Surveys. JMIR Form Res. 2022 Mar 17;6(3):e31894. doi: 10.2196/31894. PMID 35298394

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was a prospective, block randomized trial of adults undergoing elective orthopedic procedures between Jul 1-Aug 12, 2019. Objective: determine if method of digital patient engagement would impact response and completion rates. Primary outcome: response rate and total completion of PRO questionnaires. 127 participants were block randomized into receiving a mobile survey delivered as a hyperlink or responding to the same questions through an automated bidirectional texting system.
Pre-assignment Details: Patient were asked to consent via a simple SMS text message response of "yes." Only consenting patients were randomized to one of the study groups.
Period: Overall Study
Arm/Group | Treated Patients Randomized to Receive Survey | Treated Patients Randomized to Receive Text Script
Started | 63 | 64
Completed | 63 | 64
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treated Patients Randomized to Receive Survey | Treated Patients Randomized to Receive Text Script | Total
Number analyzed (Participants) | 63 | 64 | 127
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.2 (13.7) | 37.8 (14.2) | 38.5 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 26 | 54
  Male | 35 | 38 | 73
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Opioid Tablets Taken Within 28 Days
Description: We will tally number of pills taken within 28 days for each patient.
Time Frame: 28 days
Measure: Mean (Standard Deviation); unit: number of pills taken
Arm/Group | Treated Patients Randomized to Receive Survey | Treated Patients Randomized to Receive Text Script
Number analyzed (Participants) | 63 | 64
number of pills taken | 8.05 (6.02) | 11.55 (8.22)

2. Secondary Outcome: Number of Opioid Tablets Prescribed Per Procedure Encounter
Description: Tally of opioid tablets prescribed per procedure encounter before and after EMR defaults are implemented.
Time Frame: 28 days
Measure: Mean (Standard Deviation); unit: # opioid tablets prescribed / procedure
Arm/Group | Treated Patients | Treated Patients Randomized to Receive Survey | Treated Patients Randomized to Receive Text Script
Number analyzed (Participants) | 127 | 63 | 64
# opioid tablets prescribed / procedure | 7.83 (7.30) | 5.09 (5.96) | 11.03 (7.50)

3. Secondary Outcome: Perceived Ability to Manage Pain
Description: Patient's perceived ability to manage pain on a 10 point scale (10=highest, 1=lowest)
Time Frame: 28 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treated Patients Randomized to Receive Survey | Treated Patients Randomized to Receive Text Script
Number analyzed (Participants) | 63 | 64
units on a scale | 7.17 (2.90) | 6.69 (2.63)

4. Secondary Outcome: Number of Opioid Pills Remaining
Description: Tally of opioid pills left after a patient reports discontinued use.
Time Frame: 28 days
Population: Tally of opioid pills left after a patient reports discontinued use.
Measure: Mean (Standard Deviation); unit: quantity of pills remaining
Arm/Group | Treated Patients Randomized to Receive Survey | Treated Patients Randomized to Receive Text Script
Number analyzed (Participants) | 63 | 64
quantity of pills remaining | 15.62 (9.10) | 13.59 (7.12)

5. Other Pre Specified Outcome: Response Rate
Description: Number of patients who respond to automated text with a survey or bi-directional text script
Time Frame: 28 days
Population: Participant surveys/text scripts only continue to day 28 if participants stated they plan to continue taking pills. All but 1 participant discontinued taking pills by day 21. Therefore, only 1 day 28 survey was sent (the participant responded) and 0 day 28 text scripts were sent.
Measure: Count of Participants; unit: Participants
Arm/Group | Treated Patients Randomized to Receive Survey | Treated Patients Randomized to Receive Text Script
Number analyzed (Participants) | 1 | 0
Participants | 1 | 0

6. Other Pre Specified Outcome: Completion Rate
Description: Number of patients who complete the automated text survey or bi-directional text script
Time Frame: 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Treated Patients Randomized to Receive Survey | Treated Patients Randomized to Receive Text Script
Number analyzed (Participants) | 19 | 16
Participants | 18 | 9

ADVERSE EVENTS:
Time Frame: 28 days
Description: All patients surveyed were undergoing an elective outpatient orthopedic surgery where adverse events are minimal risk.
Arm/Group | Treated Patients Randomized to Receive Survey | Treated Patients Randomized to Receive Text Script
All-Cause Mortality (participants affected / at risk) | 0/63 | 0/64
Serious Adverse Events (participants affected / at risk) | 0/63 | 0/64
Other Adverse Events (participants affected / at risk) | 0/63 | 0/64

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-04): https://cdn.clinicaltrials.gov/large-docs/56/NCT03532256/Prot_SAP_000.pdf